CLINICAL TRIAL: NCT03695302
Title: Knowledge , Attitude and Practice (KAP) of Fifth Year Undergraduate Dental Students on Post Exposure Prophylaxis: An Observational Study
Brief Title: Knowledge , Attitude and Practice (KAP) of Fifth Year Undergraduate Dental Students on Post Exposure Prophylaxis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Tarek Sabry, General Practitioner, Cairo University
Other Study IDs: UCairo
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Occupational Exposure
Keywords: knowledge/attitude/practice/questionnaire/post-exposure
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaire — KAP questionnaire for fifth year undergraduate dental students.

SUMMARY:
Considering the increasing number of HIV and HBV cases, the aim of this study is to evaluate the knowledge,Attitude and practice of fifth year undergraduate dental students regarding post-exposure prophylaxis.

DETAILED DESCRIPTION:
needle stick injury is inevitable. Needle stick injury is deﬁned as penetration of a sharp instrument into the body of a healthcare professional, exposing them to high-risk body ﬂuids.

Cutaneous injuries are the most common cause of infection transmission from patient to dentist. The causes of such injuries have been reported as 37% from dental burs , 30% from syringes , 6% from orthodonticwires , 3% from suture needles, 1% from blades and 2% from other sharp instruments .

Since high-risk exposure is unavoidable, dentists should be aware of post-exposure protocols to prevent infection .

ELIGIBILITY:
Inclusion Criteria:

* All Fifth Year dental students in Faculty of Dentistry ,Cairo University at the time of the study

Exclusion Criteria:

* Refusal of participation from the students.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifth year undergraduate dental students in Faculty of Dentistry , Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge,Attitude and Practice questionnaire of fifth year undergraduate dental students on post exposure prophylaxis | 1 day
  The questionnaire will be given to students to be filled in one of their clinical sections

IPD SHARING:
Plan to Share IPD: Undecided